CLINICAL TRIAL: NCT06815328
Title: Efficacy of Shock Wave Therapy in Patients with Muscle Spasticity After a Stroke
Brief Title: Efficacy of Shock Wave Therapy in Post-Stroke Muscle Spasticity Management
Acronym: SWT-PI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Maria Blanco Diaz, Professor and Researcher, Department of Surgery and Medical-Surgical Specialties, University of Oviedo, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad de Oviedo
Record Dates: First submitted 2025-01-24; First posted 2025-02-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Spasticity; Post-stroke; Muscle Hypertonia; Neurological Disorders; Physiotherapy
Keywords: Shock Wave Therapy; Post-Stroke Spasticity; Non-Invasive Therapy; Quality of Life; Neurological physical therapy; Muscle Hypertonia Treatment
MeSH Terms: conditions — Stroke; Muscle Spasticity; Muscle Hypertonia; Nervous System Diseases | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Shock Wave Therapy (SWT) (Experimental): Participants in this arm will receive Shock Wave Therapy applied to spastic muscle groups identified during the baseline assessment. The therapy will be delivered using a focused SWT device with standardized parameters (e.g., frequency, energy level, and duration). Each session will last approximately 30 minutes and will be administered once a week for 8 weeks. The intervention targets neuromuscular modulation to reduce spasticity and improve joint mobility.
  Interventions: Other: Shock Wave Therapy (SWT)
- Conventional Therapy (Active Comparator): Participants in this arm will receive standard care for post-stroke spasticity, which may include physical therapy sessions focused on stretching, strengthening, and mobility exercises, alongside medications if prescribed (e.g., muscle relaxants). The therapy will follow current clinical guidelines and will be administered with the same frequency and duration (once a week for 8 weeks) to ensure comparability with the experimental arm.
  Interventions: Other: Active Comparator - Conventional Therapy

INTERVENTIONS:
Other: Shock Wave Therapy (SWT) — Focused SWT sessions targeting spastic muscle groups. Parameters include standardized frequency, energy level, and session duration (30 minutes per session, once weekly for 8 weeks). This therapy aims to reduce muscle spasticity, improve joint mobility, and enhance quality of life.
  Standard care consisting of physical therapy sessions (e.g., stretching, mobility exercises) and/or prescribed medications for spasticity management. The therapy follows clinical guidelines and is administered with the same frequency and duration (once weekly for 8 weeks) as the experimental intervention.
  Arms: Experimental: Shock Wave Therapy (SWT)
Other: Active Comparator - Conventional Therapy — Standard care consisting of physical therapy sessions (stretching, mobility exercises) and/or prescribed medications for spasticity management.
  Follows clinical guidelines and is administered with the same frequency and duration (once weekly for 8 weeks) as the experimental intervention.
  Arms: Conventional Therapy

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of shock wave therapy (SWT) in reducing muscle spasticity in patients who have suffered a stroke. The main questions it aims to answer are:

Does SWT reduce muscle tone and improve joint range of motion in post-stroke patients with spasticity? Does SWT improve the quality of life for these patients? What side effects, if any, occur during or after SWT? Researchers will compare SWT to conventional spasticity treatments to determine its effectiveness and potential advantages.

Participants will:

Undergo SWT sessions as part of their rehabilitation protocol over a period of 8 weeks.

Attend follow-up visits to assess muscle tone, joint mobility, and overall functional improvement.

Complete quality-of-life questionnaires to measure the therapy's impact on daily living.

DETAILED DESCRIPTION:
This study aims to assess the efficacy and safety of Shock Wave Therapy (SWT) as a non-invasive treatment for muscle spasticity in post-stroke patients. Muscle spasticity is a major complication in neurorehabilitation, affecting mobility, functionality, and quality of life. Conventional treatments, including physical therapy, oral medications, and botulinum toxin injections, have limitations such as variable efficacy, side effects, and accessibility issues. SWT has gained interest as a potential alternative, but high-quality evidence regarding its effectiveness and safety in this population remains scarce.

Study Design and Rationale The study is designed as a prospective, randomized controlled trial (RCT) comparing SWT with conventional treatment approaches. SWT delivers mechanical acoustic waves to targeted spastic muscles, aiming to reduce hypertonicity and neuromuscular dysfunction. The hypothesized mechanism of action involves neuromuscular modulation, local tissue repair promotion, and increased vascularization, which may improve muscle tone, functional mobility, and overall patient outcomes.

Participants will undergo weekly SWT sessions for 8 weeks, each lasting approximately 30 minutes. Treatment will be applied to specific muscle groups, such as the elbow flexors, wrist flexors, or calf muscles, based on baseline assessments. The frequency, intensity, and duration of SWT will follow current clinical guidelines.

The control group will receive standard care, which may include physical therapy techniques such as stretching, therapeutic exercises, and pharmacological management as per clinical indication. The study will implement a blinded assessment process, where outcome evaluators will not be aware of group allocation.

Technical Aspects of SWT Application The SWT intervention will be conducted using a focused or radial shock wave device, applying preset intensity levels tailored to spastic muscle groups. The wave frequency and energy flux density will be determined based on prior research in musculoskeletal rehabilitation. SWT will be delivered at specific treatment points over affected muscles, with adjustments as necessary according to patient response and tolerability.

Data Collection and Monitoring Data will be collected at baseline, mid-treatment (week 4), and post-treatment (week 8) using standardized clinical assessment tools. The study will also monitor for adverse events, including pain, bruising, or transient increases in spasticity, to establish a safety profile for SWT in this population.

Potential Clinical Impact If SWT demonstrates clinically significant benefits, this study could support its integration into routine post-stroke rehabilitation protocols. The findings may provide guidance for rehabilitation professionals, contribute to cost-effective management strategies, and inform clinical decision-making regarding spasticity treatment.

Ethical Compliance This study adheres to the principles of the Declaration of Helsinki and has been submitted for approval to the appropriate institutional review boards. Participants will provide written informed consent before enrollment. All collected data will be handled following confidentiality and ethical guidelines.

ELIGIBILITY:
"Inclusion Criteria":

* Adults aged 18 years or older.
* Confirmed diagnosis of stroke (ischemic or hemorrhagic) at least 6 months prior to enrollment.
* Clinically diagnosed muscle spasticity, measured by the Modified Ashworth Scale (MAS), with a score of 0 to 3.
* Stable medical condition that permits participation in the intervention.
* No significant changes in spasticity-related treatment for at least 3 months prior to the study.
* Ability to provide written informed consent to participate in the study.
* Ability to attend weekly sessions and follow-up visits as required.

"Exclusion Criteria":

* Severe spasticity or contractures unresponsive to prior treatments.
* Contraindications to Shock Wave Therapy, including:
* Local infections in the treatment area.
* Known or suspected malignancy near the treatment site.
* Severe bleeding disorders or anticoagulation therapy.
* Pregnancy.
* Neurological conditions other than stroke that could interfere with study outcomes (e.g., Parkinson's disease, multiple sclerosis).
* Recent treatments that might interfere with spasticity assessment, including:
* Injections of botulinum toxin within the past 6 months.
* Recent surgery or other interventions targeting spasticity.
* Cognitive impairment or other conditions preventing the participant from following instructions or completing study tasks.
* Severe cardiovascular, renal, or hepatic disease that might complicate therapy or participation.
* Inability to commit to follow-up visits or complete the intervention protocol due to logistical, mobility, or health-related issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Spasticity | Baseline, at 10 weeks (end of intervention), and at 12 weeks (follow-up).
  Measurement of changes in muscle tone using the Modified Ashworth Scale (MAS) from baseline to the end of the treatment period. The MAS ranges from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension).
  Units of Measure: Score from 0 to 4. Lower MAS scores indicate reduced spasticity.

SECONDARY OUTCOMES:
Change in Joint Range of Motion | Baseline, at 10 weeks (end of intervention), and at 12 weeks (follow-up).
  Measurement of changes in joint range of motion (in degrees) using a goniometer, focusing on affected joints. A higher degree value indicates better joint mobility.
Change in Quality of Life | Baseline and at 12 weeks (follow-up).
  Change in patient-reported quality of life using the Stroke Impact Scale (SIS). Units of Measure: Score from 0 to 100. Higher scores indicate better quality of life.
Grip Strength | Baseline, at 10 weeks (end of intervention), and at 12 weeks (follow-up).
  Change in grip strength, measured using a hand dynamometer. A higher grip strength value indicates better muscle function and recovery.
  Units of Measure: Kilograms (kg).
Incidence of Treatment-Related Adverse Events | Throughout the study period (12 weeks).
  Measurement of the number and nature of adverse events reported during the study, including pain, discomfort, or other side effects related to the interventions.
  Units of Measure: Count of reported adverse events.
Walking Speed | Baseline, at 10 weeks (end of intervention), and at 12 weeks (follow-up).
  Change in walking speed, assessed using the 10-Meter Walk Test (10MWT). A shorter time to complete the 10-meter distance indicates better functional mobility.
  Units of Measure: Time in seconds (s).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be shared due to privacy concerns, ethical considerations, and regulatory restrictions. Only aggregated results will be disseminated through scientific publications and presentations.